CLINICAL TRIAL: NCT06934850
Title: The Relationship Between Hand Grip Strength, Trunk Control and Functional Performance in Individuals With Mild Mental Retardation
Status: Recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burak Buğday, BURAK,BUĞDAY , PT, MSc, Lecturer in Physiotherapy and Rehabilitation, Principal Investigator, Inonu University
Other Study IDs: 2025/6862
Record Dates: First submitted 2025-03-14; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Mental Retardation
Keywords: ctional performance; trunk control,; and grip strength; ild mental retardation individua
MeSH Terms: conditions — Intellectual Disability | interventions — Hand Strength; Physical Functional Performance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mild Intellectual Disability (MID) in Children: Mild Intellectual Disability (MID) refers to a neurodevelopmental condition where a child's cognitive abilities and adaptive functioning are below average compared to peers. It typically manifests with an IQ score between 50-70 and difficulties in daily life skills, problem-solving, and academic performance.
  Interventions: Other: Hand grip strength
- Normal Development group: A typically developing child follows expected milestones in physical, cognitive, social, and emotional growth according to age. Their development occurs naturally without significant delays or disabilities.
  Interventions: Other: Hand grip strength

INTERVENTIONS:
Other: Hand grip strength — Collection Tools a) Hand Grip Force Measurement: Hand grip strength will be measured using a digital dynamometer. The measurement will be performed three times in the dominant and nondominant hand of the participant and the average value will be taken (1). b) Trunk Control Assessment: Trunk control will be assessed with the McGill core endurance test. This scale is a valid and reliable tool to objectively measure trunk stability and dynamic control levels (2). c) Motor skill assessment: Timed Up and Go Test: The Timed Up and Go Test was used to assess functional mobility and dynamic balance (3). The patient was told to get up from the chair, walk 3 meters, return and sit back in the chair. The time was recorded. Timed Stair Climbing Test: It consists of the individual climbing the stairs and returning to the starting point. The elapsed time was recorded
  Other Names: trunk control; functional performance

SUMMARY:
Scope and Limitations of the Project This project aims to examine the relationship between hand grip strength, trunk control, and functional performance in individuals with mild intellectual disability (MID). Individuals with MID face significant challenges in daily life activities and social interactions due to deficiencies in motor skills. Hand grip strength is considered a fundamental indicator of overall muscle strength and level of independence, while trunk control plays a crucial role in both postural stability and dynamic movement coordination.

The project seeks to scientifically evaluate the physical and functional parameters of these individuals and highlight the impact of motor control on daily living activities. The study is limited to individuals aged 12-18, including those with intellectual disabilities attending rehabilitation centers and healthy individuals visiting hospitals. While this limitation allows for a focused examination of the needs of a specific group, it may also restrict the generalizability of the findings to the broader population.

DETAILED DESCRIPTION:
Purpose of the Study The aim of this study is to determine the relationship between hand grip strength, trunk control, and functional performance in individuals with mild intellectual disability. In this regard, the study aims to examine the physical factors affecting motor control and functional independence in these individuals. By revealing the impact of hand grip strength on trunk stability and overall functional capacity, the study seeks to contribute to the development of specialized rehabilitation programs for these individuals.

Research Question Is there a significant relationship between hand grip strength, trunk control, and functional performance in individuals with mild intellectual disability?

Hypotheses H0 (Null Hypothesis): There is no relationship between hand grip strength, trunk control, and functional performance in individuals with mild intellectual disability.

H1 (Research Hypothesis): There is a positive and significant relationship between hand grip strength, trunk control, and functional performance in individuals with mild intellectual disability.

Objectives of the Study To measure hand grip strength in individuals with mild intellectual disability and compare it with the normal population.

To determine trunk control levels in these individuals and examine its relationship with hand grip strength.

To assess functional performance (level of participation in daily living activities) and determine its correlation with hand grip strength.

To identify the key physical parameters that should be emphasized in rehabilitation programs based on the findings.

Significance of the Study Motor control and functional limitations commonly observed in individuals with mild intellectual disability can negatively affect their participation in daily life activities. Hand grip strength is a crucial indicator of both overall muscle strength and independence in daily activities. The results of this study could provide a scientific basis for developing physical rehabilitation and occupational therapy approaches tailored for individuals with special needs. Additionally, this research aims to highlight the importance of targeted interventions to improve the quality of life for these individuals.

By focusing on a specific population, this study seeks to provide practical and applicable findings and serve as a reference for similar studies conducted in specialized centers.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild mental retardation
* Individuals aged between 12 and 18 years
* Sufficient physical ability to perform hand grip strength measurements

Exclusion Criteria:

* Impaired trunk control due to an orthopedic or neurological disorder
* Psychological or physical conditions that prevent active participation in the assessments
* Mental illnesses or physical disorders in otherwise healthy individuals that may affect measurement outcomes

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This research is designed to examine the relationship between hand grip strength, trunk control and functional performance in individuals with mild mental retardation. Data collection will be carried out in accordance with ethical rules from rehabilitation and hospitalized individuals.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-26 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Mean Hand Grip Strength in kilograms (kg) | Baseline (Day 0) and Week 8
  Hand grip strength will be measured using a standard Jamar dynamometer in a seated position, with the elbow flexed at 90 degrees. The best of three consecutive trials for each hand will be recorded and averaged.
  Unit of Measure: kilograms (kg)
Trunk Control Test Score (0-100 points) | Measured at baseline (Day 0) and at the end of the 8-week intervention period (Week 8)
  Trunk control will be evaluated using the Trunk Control Test (TCT), which assesses four functional movements: rolling to the weak side, rolling to the strong side, sitting up from lying down, and maintaining a sitting position. Each task is scored, and total scores range from 0 to 100.
  Unit of Measure: points (0-100)
Total Functional Independence Measure (FIM) Score | Baseline (Day 0) and Week 8
  Functional performance will be assessed using the Functional Independence Measure (FIM), which evaluates self-care, mobility, communication, and social cognition. Scores range from 18 to 126, with higher scores reflecting greater independence.
  Unit of Measure: points (18-126)

CONTACTS AND LOCATIONS:
Locations (1):
- Malatya Training and Research Hospital, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Hand grip strength as a proposed new vital sign of health: a narrative review of evidences — https://pubmed.ncbi.nlm.nih.gov/38195493/
- Available data/document: Clinical Study Report — https://etik.inonu.edu.tr/panel/index